CLINICAL TRIAL: NCT04750278
Title: A Phase 2/3, Randomized, Double Blind, Placebo Controlled, Multicenter Study to Evaluate the Efficacy and Safety of FP-025 in Patients With Severe to Critical COVID 19 With Associated Acute Respiratory Distress Syndrome (ARDS)
Brief Title: A Phase 2/3 Study to Evaluate FP-025 in Patients With Severe to Critical COVID 19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study stopped at interim analysis point, due to lack of study subjects to recruit.
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FP02C-20-001
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2022-08

CONDITIONS: Severe to Critical COVID 19 With Associated ARDS
MeSH Terms: interventions — FP-025; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of FP-025 in Patients With Severe to Critical COVID 19 With Associated Acute Respiratory Distress Syndrome (ARDS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FP-025 100 mg (Experimental): Low dose for patient treatment.
  Interventions: Drug: FP-025 100 mg
- FP-025 300 mg (Experimental): High dose for patient treatment.
  Interventions: Drug: FP-025 300 mg
- Placebo (Placebo Comparator): Dose without any study drug, to make it a controlled study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FP-025 100 mg — FP-025 100 mg BID
  Other Names: Active
  Arms: FP-025 100 mg
Drug: FP-025 300 mg — FP-025 300 mg BID
  Other Names: Active
  Arms: FP-025 300 mg
Drug: Placebo — Placebo BID
  Other Names: Non-Active
  Arms: Placebo

SUMMARY:
This is a Phase 2/3, randomized, double blind, placebo controlled, multicenter study to evaluate the efficacy and safety of FP-025 in adult patients with severe to critical COVID 19 with associated ARDS.

DETAILED DESCRIPTION:
This is a Phase 2/3, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of FP-025 in adult patients with severe to critical COVID-19 with associated ARDS. The patients in each phase (Phase 2 and Phase 3) will be analyzed separately. Each phase will consist of a Screening Visit, Treatment Period, and Follow-Up Period for a total study duration of approximately 60 days.

Phase 2: After eligibility is confirmed, approximately 90 patients will be randomized in a 1:1:1 ratio to receive FP-025 100 mg twice daily (BID), FP-025 300 mg BID, or placebo BID for 28 days. During Phase 2, randomized patients will be stratified by the use of invasive mechanical ventilation at the time of randomization (yes or no). At least one-third of patients should be on invasive mechanical ventilation to ensure that treatment benefits can be assessed for patients at different severity levels.

Patients with Grade 3 to Grade 4 heart failure, Stage 3 or greater chronic obstructive pulmonary disease, persistent asthma, and mild liver disease (ie, Child-Pugh Class A) will not be excluded from the study. The independent Data Monitoring Committee (iDMC) will independently monitor safety of the entire population and in different subgroups and may make recommendations as it deems appropriate. During Phase 2, no limitation in enrollment of subgroups is expected, unless clear safety signals arise in those subgroups during iDMC reviews.

The reason for hospital admission, the standard of care followed for each patient and center, and whether any care decisions were based on resource limitations will be clearly documented for all patients beginning on Day 1 (Visit 2). All patients will be allowed to receive standard of care and/or emergency use authorization (EUA) medications and treatment for COVID-19; however, the study drug should be discontinued for other non-standard of care concomitant medications used with the intent of directly treating COVID-19 unless there is prior Medical Monitor or Sponsor approval for the patient to remain on the study drug. If the use of concomitant medications necessitates study drug discontinuation, the patient should be encouraged to remain in the study and to follow-up for key study visits (Day 28 and Day 60) but will not be required to attend every study visit. If the patient withdraws, he/she should complete the Early Termination Visit.

Standard of care procedures for mechanical ventilation (eg, low tidal volume protective mechanical ventilation) and standard of care procedures for weaning from mechanical ventilation will be followed.

Study drug administration will begin on Day 1 (Visit 2) following randomization. All patients will receive standard of care and/or EUA treatment for COVID-19 in addition to the study drug. Patients will continue study drug treatment BID through Day 27 and take 1 dose on Day 28. If a patient is discharged from the hospital prior to Day 28, he/she will continue treatment as an outpatient at home with his/her assigned treatment (FP-025 100 mg BID, FP-025 300 mg BID, or placebo BID) until Day 28. Dosing instructions will be provided prior to discharge. Although treatment will be identical for inpatients and outpatients, patients discharged from the hospital will follow a different Schedule of Procedures, characterized by telemedicine (or telephone, if sites and/or patients do not have video capability) visits. The End of Treatment (EOT) Visit on Day 28 will be identical for all patients (with the exception of the arterial oxygen partial pressure [PaO2]/fractional inspired oxygen [FiO2] ratio, performed only in patients on invasive or non-invasive ventilation) and will include a high-resolution, non-contrast CT scan, in addition to other assessments.

After treatment is completed, all patients will undergo 2 follow-up assessments during the Follow-Up Period. The first follow-up will be a telephone visit on Day 45 to assess concomitant medications, adverse events (AEs), and the NIAID 8-point ordinal scale for COVID-19 and hospitalization outcomes score. The second follow-up will be an in-person visit on Day 60 and will include a high-resolution, non-contrast CT scan and pulmonary function tests, in addition to other assessments.

An iDMC will convene to oversee safety and efficacy assessments during and after the Phase 2 study. No formal statistical testing will be conducted. In addition, when all patients in the Phase 2 study have completed the EOT Visit on Day 28, a primary analysis will be conducted by an independent statistician and reviewed by the iDMC. This is the point at which the study was terminated, due to lack of further eligible patients.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing to provide informed consent (or has a legally authorized representative [LAR] willing to provide informed consent) and is willing and able (or has an LAR willing and able) to comply with the protocol required therapy, monitoring, and follow-up;
2. Is a male or female aged ≥ 18 years;
3. Has a COVID-19 diagnosis confirmed by a documented, positive severe acute respiratory syndrome (SARS) CoV-2 reverse transcriptase polymerase chain reaction test (or equivalent test) immediately prior to or during the current hospitalization;
4. Is hospitalized with severe to critical COVID 19 within a 72-hour period prior to the Screening Visit and meeting the following characteristics:

   * Diagnosed with ARDS based on the Berlin criteria as follows:

     * Respiratory symptoms developed within 1 week of a known clinical insult or new or worsening respiratory symptoms developed during the past week;
     * Chest radiograph or computed tomography scan shows bilateral opacities not fully explained by pleural effusions, lobar or lung collapse, or pulmonary nodules; and
     * Respiratory failure is not fully explained by cardiac failure or fluid overload; and
   * Requiring at least 1 of the following:

     * Endotracheal intubation and mechanical ventilation;
     * Oxygen delivered by high flow nasal cannula (heated, humidified oxygen delivered via reinforced nasal cannula at flow rates > 20 L/minute with a fraction of delivered oxygen ≥ 0.5);
     * Non invasive positive pressure ventilation; or
     * Clinical diagnosis of respiratory failure (ie, the clinical need for 1 of the preceding therapies, but preceding therapies are unable to be administered in the setting of resource limitations);
5. If female, is post-menopausal for at least 1 year, surgically sterile (documented by medical record), or a woman of childbearing potential (WCBP) who agrees to use a highly effective method of birth control (ie, method with a failure rate < 1% per year) from enrollment until 30 days following the last dose of study drug. Highly effective methods of birth control are defined as follows: complete sexual abstinence, intrauterine device, intrauterine hormone-releasing system, progestogen-only hormonal contraception (implant, injectable, or oral), and combined (estrogen and progestogen) contraception (oral, intravaginal, or transdermal);
6. If a WCBP, must have a negative serum human chorionic gonadotropin pregnancy test at the Screening Visit, and must agree to monthly urine pregnancy tests during the study; and
7. If male, must be surgically sterile for at least 1 year prior to the Screening Visit (documented by medical record), or must agree to use a double barrier approach (eg, condoms with spermicide) during sexual intercourse between the Screening Visit and at least 90 days after administration of the last dose of study drug. Male patients must ensure that non pregnant female partners of childbearing potential comply with the contraception requirements in Inclusion Criterion 5.

Exclusion Criteria:

1. Is not expected to survive more than 24 hours;
2. Is on extracorporeal membrane oxygenation (ECMO) at the Screening Visit;
3. Has an underlying clinical condition where, in the opinion of the Investigator, it would be extremely unlikely that the patient would come off ventilation (eg, motor neuron disease, Duchenne muscular dystrophy, or rapidly progressive pulmonary fibrosis);
4. Has a known history of idiopathic pulmonary fibrosis or interstitial lung disease as defined by the American Thoracic Society 2018 guidelines;
5. Has known active tuberculosis (TB), a history of incompletely treated TB, and/or suspected or known extrapulmonary TB;
6. Has Child Pugh Class B or C active liver disease or an alanine aminotransferase or aspartate aminotransferase level > 4 x the upper limit of normal at the Screening Visit;
7. Has moderate to severe renal insufficiency, defined as an estimated glomerular filtration rate (eGFR) ≤ 30 mL/min/1.73 m2, at the Screening Visit or requires hemodialysis;
8. Has a malignant tumor (excluding a malignant tumor cured with no recurrence in the past 5 years, completely resected basal cell and squamous cell carcinoma of skin, and/or completely resected carcinoma in situ of any type);
9. Has an uncontrolled systemic or local autoimmune or inflammatory disease besides COVID 19;
10. Has evidence of an active concurrent non COVID 19 pneumonia (requiring additional antimicrobial treatment) caused by a known or suspected bacterial pathogen, respiratory syncytial virus (RSV), influenza virus, SARS CoV 1, Middle East respiratory syndrome CoV, aspergillus, mucormycosis causing fungi, or other pulmonary pathogen(s);

    Note: A viral respiratory panel will be administered at the Screening Visit to determine eligibility. At a minimum, the panel will evaluate for RSV, influenza A, and influenza B.
11. Has received any other investigational therapeutic products within 4 weeks or 5 half-lives, whichever is longer, prior to randomization;
12. Has a known history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection;
13. Has a known serious allergic reaction or hypersensitivity to any components of FP-025;
14. Is pregnant or breastfeeding;
15. Has a history of drug or alcohol abuse within the past 2 years;
16. Is currently on another systemic immunomodulatory therapy that is not considered standard of care treatment for COVID 19 (eg, calcineurin inhibitor, hydroxychloroquine, anti cytokine therapy, or Janus kinase inhibitor); or Note: Corticosteroids, including dexamethasone, in doses used for standard of care treatment for COVID 19 are allowed.

    Note: Corticosteroids that are being used for other indications are also allowed as long as the daily prednisone (or other corticosteroid equivalent) dose is ≤ 10 mg. Inhaled corticosteroids and nasal corticosteroids are also acceptable.

    Note: As therapies for COVID-19 are rapidly evolving, other medications that may be considered standard of care can be considered with prior approval from the Sponsor or Medical Monitor.
17. Has any other condition that, in the opinion of the Investigator, could interfere with (or for which the treatment might interfere with) the conduct of the study or interpretation of the study results or that would place the patient at undue risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shelby, Ph.D., Study Director — Sr. Vice President Clinical Development
Locations (8):
- United States (8):
  - Velocity Chula Vista, Chula Vista, California
  - Velocity San Diego, La Mesa, California
  - Shady Grove Medical Center, Rockville, Maryland
  - University of Nevada, Las Vegas (UNLV) School of Medicine, Las Vegas, Nevada
  - Trinity Health Center, Minto, North Dakota
  - Legacy Health, Portland, Oregon
  - Houston Methodist, Houston, Texas
  - United Medical Memorial Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FP-025 300 mg: High dose for patient treatment.
  FP-025 300 mg: FP-025 300 mg BID
  30 subjects
- FP-025 100 mg: Low dose for patient treatment.
  FP-025 100 mg: FP-025 100 mg BID
  29 subjects
- Placebo: Dose without any study drug, to make it a controlled study.
  Placebo: Placebo BID
  31 subjects
Period: Overall Study
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Started | 30 | 29 | 31
Completed D28 Visit | 16 | 16 | 18
Completed | 15 | 13 | 15
Not Completed | 15 | 16 | 16
Not completed — Death | 9 | 10 | 10
Not completed — Withdrawal by Subject | 4 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Legally Authorized Representative | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Transfer to Outside Facility | 0 | 2 | 1
Not completed — Staff Inadvertently Failed to Follow up with Subject Visits | 0 | 1 | 0
Not completed — Patient Hospitalized Secondary to Unrelated SAE and Did Not Have Study Medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients with COVID-19 acute respiratory distress syndrome who met the inclusion criteria of the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | FP-025 100 mg | FP-025 300 mg | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 31 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 26 | 71
  >=65 years | 5 | 9 | 5 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 5 | 29
  Male | 17 | 18 | 26 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 3 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 3 | 6
  White | 19 | 19 | 14 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 10 | 22
Number of patients on mechanical ventilation [Count of Participants; unit: Participants] | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Alive and Not Requiring Non-invasive or Invasive Ventilation
Description: Percentage of patients alive and not requiring non-invasive or invasive ventilation at Day 28
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants
  Meeting the primary efficacy endpoint | 15 | 10 | 18
  Not meeting the primary efficacy endpoint | 15 | 19 | 13

2. Secondary Outcome: Percentage of Patients on Invasive Mechanical Ventilation
Description: Percentage of patients on invasive mechanical ventilation at Day 28
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants
  Percentage of patients on invasive mechanical ventilation at Day 28 | 10 | 14 | 11
  Percentage of patients not on invasive mechanical ventilation at Day 28 | 20 | 15 | 20

3. Secondary Outcome: Percentage of Patients Alive
Description: Percentage of patients who are alive at the time of the assessment, day 28.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants
  Percentage of patients alive at Day 28 | 21 | 19 | 22
  Percentage of patients not alive at Day 28 | 9 | 10 | 9

4. Secondary Outcome: Percentage of Patients Alive and Not Requiring Non-invasive or Invasive Ventilation
Description: (ie, not receiving high flow nasal cannula, non-invasive positive pressure ventilation, invasive mechanical ventilation, or ECMO)
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants | 12 | 10 | 13

5. Secondary Outcome: Percentage of Patients on Invasive Mechanical Ventilation
Description: Percentage of patients receiving high flow nasal cannula, non-invasive positive pressure ventilation, invasive mechanical ventilation, or ECMO at day 60
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants
  Percentage of patients on invasive mechanical ventilation at Day 60 | 10 | 13 | 11
  Percentage of patients not on invasive mechanical ventilation at Day 60 | 20 | 16 | 20

6. Secondary Outcome: Percentage of Patients Alive
Description: Percentage of patients who continue to be alive at day 60.
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants
  Percentage of patients alive at Day 60 | 21 | 19 | 21
  Percentage of patients not alive at Day 60 | 9 | 10 | 10

7. Other Pre Specified Outcome: Quantitative Assessment of Lung Fibrosis
Description: Percentage of patients having lung fibrosis using high resolution, non-contrast CT scan, at days 28 and 60
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percentage of Patients Who Were Randomized on Invasive Mechanical Ventilation Who Are Free of Invasive Mechanical Ventilation
Description: Percentage of patients at days 28 and 60 who improved to breathing on their own, after having been on mechanical ventilation at some point during their treatment.
Time Frame: Day 28 and at Day 60
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Ventilator Free Days (ie, Days Free of Invasive Mechanical Ventilation)
Description: Number of days (out of 28 and 60, respectively) that patient is off of mechanical ventilation.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of ICU Free Days
Description: Number of days (out of 28 and 60, respectively) that the patient is not in the ICU
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Days in the Hospital
Description: Number of days (out of 28 and 60, respectively) that the patient is hospitalized.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change From Baseline in Peripheral Capillary Oxygen Saturation (SpO2)
Description: The number of percentage points the patient has changed in peripheral capillary oxygen saturation (SpO2) at days 28 and 60.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline in Arterial Oxygen Partial Pressure (PaO2)/Fractional Inspired Oxygen (FiO2) Ratio
Description: Change from baseline, at days 28 and 60, in arterial oxygen partial pressure .(PaO2)/fractional inspired oxygen (FiO2) ratio.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Percentage of Patients Alive and Not Hospitalized
Description: Percentage of patients at day 28 and day 60 who are alive and not hospitalized.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Percentage of Patients With Disease Progression
Description: (defined as a ≥ 2 point decrease in the NIAID 8 point ordinal scale score or death)
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Percentage of Patients Who Improve by ≥ 2 Points on the NIAID 8 Point Ordinal Scale Scores
Description: Percentage of patients who improve by ≥ 2 points on the NIAID 8 point ordinal scale scores at Day 28 and Day 60
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Pulmonary Function Test
Description: Measured by Forced Expiratory Volume in 1 second (FEV1) /Forced Vital Capacity (FVC) at Day 28 and Day 60
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change From Baseline in eGFR
Description: Change from baseline in eGFR at day 28 and day 60.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change From Baseline in Blood Urea Nitrogen
Description: Change .from baseline in blood urea nitrogen at day 28 and day 60
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change From Baseline in Serum Creatinine
Description: Change from baseline in serum creatinine at day 28 and day 60.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change From Baseline in HRQoL as Measured by the EQ 5D 5L
Description: Change from baseline in HRQoL as measured by the EQ 5D 5L at day 28 and day 60.
Time Frame: Day 28 and Day 60
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 60 days
Description: Participants at Risk were considered to be participants in the safety population of the study. The safety population is defined as any participant who received at least one dose of study drug or placebo. This differs from the intent to treat population which is defined as any participant who was randomized to receive study drug or placebo. One (1) patient in the 100 mg group and one (1) patient in the placebo group did not receive study drug or placebo. Both patients withdrew consent.
Groups:
- FP-025 100 mg: Low dose for patient treatment.
  FP-025 100 mg: FP-025 100 mg BID
  28 subjects
- Placebo: Dose without any study drug, to make it a controlled study.
  Placebo: Placebo BID
  30 subjects
Arm/Group | FP-025 300 mg | FP-025 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 9/30 | 10/29 | 10/31
Serious Adverse Events (participants affected / at risk) | 11/30 | 12/28 | 11/30
Other Adverse Events (participants affected / at risk) | 17/30 | 21/28 | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-025 300 mg (N=30) | FP-025 100 mg (N=28) | Placebo (N=30)
Infections and infestations (Infections and infestations) | 3 (3) | 4 (4) | 5 (5)
Cardiac Disorders (Cardiac disorders) | 3 (3) | 5 (6) | 3 (6)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (2)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FP-025 300 mg (N=30) | FP-025 100 mg (N=28) | Placebo (N=30)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (10) | 5 (5)
Infections and infestations (Infections and infestations) | 5 (6) | 7 (13) | 7 (9)
Cardiac disorders (Cardiac disorders) | 5 (6) | 6 (9) | 5 (9)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (8) | 3 (4) | 4 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (4) | 4 (5) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 3 (3) | 3 (3)
Psychiatric disorders (Psychiatric disorders) | 2 (2) | 6 (6) | 0 (0)
Vascular disorders (Vascular disorders) | 2 (6) | 4 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT04750278/Prot_SAP_000.pdf